CLINICAL TRIAL: NCT02705053
Title: At Home Study of a Zone-Model Predictive Control (MPC) Controller and a Health Monitoring System (HMS) With the Diabetes Assistant (DiAs) System and Run-to-Run Adaptation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Harvard University (Other); University of California, Santa Barbara (Other); Mayo Clinic (Other); University of Virginia (Other); University of Padova (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G150063_2
Record Dates: First submitted 2016-02-25; First posted 2016-03-10 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 1; Artificial Pancreas; Autoimmune Diseases; Diabetes Mellitus; Hyperglycemia; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases; Diabetes Mellitus; Hyperglycemia; Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sensor-Augmented Pump Open-Loop Care (Week 2) (Active Comparator): The subjects' Sensor-Augmented Pump Open-Loop Care for the second week of the study before any adjustments to pump settings, using a CGM and Insulin Pump.
  Interventions: Device: CGM and Insulin Pump
- Closed-Loop Control System with Zone MPC and HMS (Experimental): The artificial pancreas system will be allowed to employ its Model Predictive Control algorithm to make decisions about insulin delivery based on CGM glucose levels. The Health Monitoring System algorithm uses the same CGM data as the MPC control algorithm but utilizes a separate algorithm for trending and predictions of future glucose values. Using a redundant and independent algorithm is an important safety feature of the overall AP device. Algorithmic adjustment of carbohydrate ratios prior to closed-loop initiation, and continued basal rate and carbohydrate ratio algorithmic optimization during closed-loop use will occur.
  Interventions: Device: Closed-Loop Control System

INTERVENTIONS:
Device: CGM and Insulin Pump — Dexcom G4 Platinum CGM with Share AP Receiver Roche Accu-Chek insulin pump.
  Arms: Sensor-Augmented Pump Open-Loop Care (Week 2)
Device: Closed-Loop Control System — The devices that will be used in the Closed-Loop Control System include the following components:
  DiAs - a smart-phone medical platform; Dexcom G4 Platinum connected to DiAs via Bluetooth CGM receiver; Roche Accu-Chek insulin pump connected to DiAs via wireless Bluetooth; Remote Monitoring Server connected to DiAs via 3G or local Wi-Fi network, and Zone-MPC and HMS algorithms running on DiAs (MPC and HMS)
  Arms: Closed-Loop Control System with Zone MPC and HMS

SUMMARY:
This clinical trial is a study to assess the performance of an automated glucose control system (Artificial Pancreas, AP) device in home settings for subjects with type 1 diabetes. Specifically, the investigators will test zone model predictive control AP that will be enhanced by run-to-run optimizations of basal rates (BR) and insulin to carbohydrate ratios (CR).

DETAILED DESCRIPTION:
This clinical trial is a study to assess the performance of an automated glucose control system (Artificial Pancreas, AP) device in home settings for subjects with type 1 diabetes. Specifically, the investigators will test zone model predictive control AP that will be enhanced by run-to-run optimizations of basal rates (BR) and insulin to carbohydrate ratios (CR). This protocol builds on the investigators previously validated Zone-MPC and Health Monitoring System (HMS) algorithms (ClinicalTrials.gov: NCT01929798) integrated into the Diabetes Assistant (DiAs) system (ClinicalTrials.gov: NCT02463682). The same AP system used in NCT02463682 will now be used with algorithmic adjustment of CR's prior to closed-loop initiation, and continued BR and CR algorithmic optimization during closed-loop use for a longer duration.

The system will be evaluated on up to 12 subjects per site (n=36 subjects) for 15 weeks at 3 different sites (William Sansum Diabetes Center, University of Virginia, and Mayo Clinic, Rochester, MN).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least 1 year and an insulin pump for at least 6 months
* Willing to wear the study CGM device for the duration of the study
* Age ≥21 to <65 years
* HbA1c <10.0%; if HbA1c <6.0% then total daily insulin must be ≥0.5 U/kg
* For females, not currently known to be pregnant. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study.
* Demonstration of proper mental status and cognition for the study
* Currently using insulin-to-carbohydrate ratio to calculate meal bolus sizes
* Hypoglycemia awareness as demonstrated by a Clarke Hypoglycemia Unawareness score of 2 or lower
* Access to internet and cell phone service at home, and a computer for downloading device data
* Availability of care partner committed to participating in training activities, knowledgeable at all times of the participant's location, and being available to provide assistance when system is being used at night
* Commitment to maintaining uninterrupted availability via cell phone and avoiding any overnight travel for the duration the period using the closed-loop system
* An understanding of and willingness to follow the protocol and sign the informed consent

Exclusion Criteria:

* Admission for diabetic ketoacidosis in the 12 months prior to enrollment
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
* History of a seizure disorder (except hypoglycemic seizure), unless written clearance is received from a neurologist
* Coronary artery disease or heart failure, unless written clearance is received from a cardiologist
* History of cardiac arrhythmia (except for benign premature atrial contractions and benign premature ventricular contractions which are permitted)
* Cystic fibrosis
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

  1. Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver (i.e., parent or guardian)
  2. Presence of a known adrenal disorder
  3. Abnormal liver function test results (Transaminase >2 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function
  4. Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2); testing required for subjects with diabetes duration of greater than 5 years post onset of puberty
  5. Active gastroparesis
  6. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
  7. Uncontrolled thyroid disease (TSH undetectable or >10 mlU/L); testing required within three months prior to admission for subjects with a goiter or who are on thyroid hormone replacement, and within one year otherwise
  8. Abuse of alcohol or recreational drugs
  9. Infectious process not anticipated to resolve prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis)
* A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol
* Current use of the following drugs and supplements:

  1. Acetaminophen
  2. Beta blockers
  3. Oral or injectable glucocorticoids
  4. Any other medication that the investigator believes is a contraindication to the subject's participation

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) (%) from baseline (week 2) to end of week 15 (end of study), with A1c measured at weeks 7 and 11 as well for repeated measures. | 13 Weeks
  The primary endpoint is change in HbA1c from baseline (end of week 2) to end of week 15 (end of study). HbA1c will be measured at weeks 7 and 11 as well following each adaptation period, so the overall design of the study includes 4 repeated measures and a baseline-end of study contrast.

SECONDARY OUTCOMES:
Time within the target range for glucose 70-180 mg/dl overall | 1 week
  Time within the target range for glucose 70-180 mg/dl overall, compared between sensor-augmented pump use (open loop care, week 2) and adapted closed-loop control (final week of each month) to determine the feasibility of long-term system use.
Time within the tight target range for glucose 80-140 mg/dl overnight | 1 week
  Time within the tight target range for glucose 80-140 mg/dl overnight, compared between sensor-augmented pump use (open loop care, week 2) and adapted closed-loop control (final week of each month) to determine the feasibility of long-term system use.
Time within the target range for glucose 70-150 mg/dl postprandial within 5 hours following meals | 1 week
  Time within the target range for glucose 70-150 mg/dl postprandial within 5 hours following meals, compared between sensor-augmented pump use (open loop care, week 2) and adapted closed-loop control (final week of each month) to determine the feasibility of long-term system use.
Markers of hypo- and hyperglycemia | 1 week
  Markers of hypo- and hyperglycemia, compared between sensor-augmented pump use (open loop care, week 2) and adapted closed-loop control (final week of each month) to determine the feasibility of long-term system use. These markers include LBGI (Low blood glucose index) and HBGI (High blood glucose index.
Insulin Doses Given | 1 week
  Change in insulin doses given, compared between sensor-augmented pump use (open loop care, week 2) and adapted closed-loop control (final week of each month) to determine the feasibility of long-term system use.
Treatments for hypoglycemia | 1 week
  Treatments for hypoglycemia between the open and closed-loop phases of the study, compared between sensor-augmented pump use (open loop care, week 2) and adapted closed-loop control (final week of each month) to determine the feasibility of long-term system use.
Number of alerts given by the HMS to prevent hypoglycemia | 12 weeks
  Number of alerts given by the HMS to prevent hypoglycemia during closed-Loop control.
Outside interventions needed. | 12 weeks
  Outside interventions needed to aid with treatment during closed-Loop control.
Failure analysis of the devices/connectivity issues that may occur (# disconnects and device restarts). | 12 weeks
  Failure analysis of the devices/connectivity issues that may occur during closed-Loop control. This includes number of CGM communication losses with 3 or more missed points, and number of times the entire system required a restart
Time with glucose ≤ 70 mg/dL, overall | 1 week
  Time with glucose ≤ 70 mg/dL, compared between sensor-augmented pump use (open loop care, week 2) and adapted closed-loop control (final week of each month) to determine the feasibility of long-term system use.

CONTACTS AND LOCATIONS:
Overall Officials: Francis J Doyle III, PhD, Principal Investigator — Harvard University; Eyal Dassau, PhD, Principal Investigator — Harvard University; Jordan E Pinsker, MD, Principal Investigator — Sansum Diabetes Research Institute; Ananda Basu, MD, Principal Investigator — Mayo Clinic, Rochester, MN; Yogish Kudva, MD, Principal Investigator — Mayo Clinic, Rochester, MN; Boris Kovatchev, PhD, Principal Investigator — University of Virginia; Sue Brown, MD, Principal Investigator — University of Virginia; Stephen Patek, PhD, Principal Investigator — University of Virginia; Claudio Cobelli, PhD, Principal Investigator — University of Padova
Locations (3):
- United States (3):
  - William Sansum Diabetes Center, Santa Barbara, California
  - Mayo Clinic, Rochester, Minnesota
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dassau E, Pinsker JE, Kudva YC, Brown SA, Gondhalekar R, Dalla Man C, Patek S, Schiavon M, Dadlani V, Dasanayake I, Church MM, Carter RE, Bevier WC, Huyett LM, Hughes J, Anderson S, Lv D, Schertz E, Emory E, McCrady-Spitzer SK, Jean T, Bradley PK, Hinshaw L, Laguna Sanz AJ, Basu A, Kovatchev B, Cobelli C, Doyle FJ 3rd. Twelve-Week 24/7 Ambulatory Artificial Pancreas With Weekly Adaptation of Insulin Delivery Settings: Effect on Hemoglobin A1c and Hypoglycemia. Diabetes Care. 2017 Dec;40(12):1719-1726. doi: 10.2337/dc17-1188. Epub 2017 Oct 13. PMID 29030383